CLINICAL TRIAL: NCT01589003
Title: An Intervention Study to Consider the Impact of Milk-products Differing in Their Glycaemic Properties on the Behaviour of Infants.
Brief Title: The Impact of Milk-products Differing in Their Glycaemic Properties on the Behaviour of Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Geok Lin Khor (Other)
Collaborators: Fonterra Research Centre (Industry)
Responsible Party: Sponsor-Investigator, Geok Lin Khor, Professor Khor Geok Lin, IMU University, Malaysia
Organization: IMU University, Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: Acute01
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Mood Behaviour; Cognitive Function
Keywords: low GI milk mood behaviour cognitive function children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low GI group (Active Comparator): Low Glycaemic index growing up milk
  Interventions: Other: Low Glycaemic index growing up milk
- High GI group (Other): Hi Glycaemic index growing up milk
  Interventions: Other: High GI growing up milk

INTERVENTIONS:
Other: Low Glycaemic index growing up milk — Low Glycaemic index growing up milk
  Arms: Low GI group
Other: High GI growing up milk — High glycaemic index growing up milk
  Arms: High GI group

SUMMARY:
The current study proposes to investigate the impact of a low glycaemic index (GI), fortified toddlers milkpowder on mood, behaviour and cognitive function in young children.

DETAILED DESCRIPTION:
The current study proposes to investigate the impact of a low GI, fortified toddlers milkpowder on mood, behaviour and cognitive function in young children. In choosing the tests it should be remembered that the investigators looking for short-term changes in functioning, such as the ability to sustain attention or improved mood. As such the investigators are not looking for measures of general cognitive functioning, stage of development or general behaviour but rather measures that are capable of monitoring changes from hour to hour or day to day.

ELIGIBILITY:
Inclusion Criteria:

* The sample will consist of only Malay children, an equal number of boys and girls, and whose parents have consent to the child participating in this trial.

Exclusion Criteria:

* they will be excluded if underweight (BMI for age < 2 S.D.);
* overweight (BMI for age > 2 S.D.;
* have any chronic or serious illness or are currently not feeling well / taking medication;
* have a history of allergy (particularly to milk), thyroid disease or diabetes mellitus.

Children currently part of an iron/zinc supplementation programme will be excluded as will any who are still being breast fed as there is no intention to discourage breastfeeding

Ages: 15 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-10 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
The impact of a low GI, fortified toddlers milkpowder on mood, behaviour and cognitive function in young children | 5 days
  Evaluated by Parental ratings, Tempertment mood questionnaires, Ethological description of free play, Distractability task, actiwatch, Sleep Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: David Benton, Professor, Study Chair — Swansea University; Geok Lin Khor, Professor, Principal Investigator — International Medical University Malaysia; Peter Mitchell, Professor, Study Chair — University of Nottingham Malaysia Campus; Dr Shamsul Haque, PhD, Study Chair — Monash University Sunway Campus Malaysia; Snigdha Misra, PhD, Study Chair — International Medical University Malaysia
Locations (1):
- Childcare centres, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Misra S, Khor GL, Mitchell P, Haque S, Benton D. A pilot study to determine the short-term effects of milk with differing glycaemic properties on sleep among toddlers: a randomised controlled trial. BMC Pediatr. 2015 Jul 15;15:79. doi: 10.1186/s12887-015-0393-9. PMID 26174581